CLINICAL TRIAL: NCT00002680
Title: Phase II Trial of Sequential High-Dose Alkylating Agents in Metastatic Breast Cancer
Brief Title: Sequential High-Dose Chemotherapy and Stem Cell Transplantation in Treating Patients With Chemotherapy-Sensitive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000064338; YALE-HIC-7372; NCI-V95-0721
Record Dates: First submitted 1999-11-01; First posted 2004-04-29 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2009-08

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; Cyclophosphamide; Megestrol Acetate; Melphalan; Tamoxifen; Thiotepa; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
Drug: megestrol acetate
Drug: melphalan
Drug: tamoxifen citrate
Drug: thiotepa
Procedure: conventional surgery
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of sequential high-dose chemotherapy followed by peripheral stem cell transplantation in treating patients with metastatic breast cancer that is responding to chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility and efficacy of sequential high-dose cyclophosphamide, melphalan, and thiotepa plus autologous peripheral blood stem cell rescue in patients with metastatic breast cancer with ongoing objective response to prior induction chemotherapy.

OUTLINE: Patients receive sequential therapy beginning with regimen A. Regimen A: Patients receive cyclophosphamide IV over 1 hour every 6 hours or more for 4 doses within 36 hours. Patients receive filgrastim (G-CSF) subcutaneously (SC) daily beginning 2 days after completion of cyclophosphamide and continuing until autologous peripheral blood stem cells (PBSC) are harvested. Regimen B: Beginning at least 3 weeks after initiation of regimen A, patients receive melphalan IV on days 1 and 2. Beginning on day 4, a portion of the PBSC are reinfused. Patients receive G-CSF SC daily beginning on day 4 and continuing until at least day 10. Regimen C: Beginning at least 3 weeks after initiation of regimen B, patients receive thiotepa IV over 2 hours on days 1 and 2. Beginning on day 5, the remaining PBSC are reinfused. Patients receive G-CSF SC daily beginning on day 5 and continuing until blood counts recover. During regimens A, B, and C, G-CSF must be discontinued at least 2 days before administration of any chemotherapy. Regimen D: After recovery from chemotherapy, patients with hormone receptor-positive tumors and no prior refractoriness to hormonal therapies receive oral tamoxifen daily, while patients with prior failure on tamoxifen receive oral megestrol 4 times daily. Patients undergo irradiation to sites of prior cutaneous, nodal, bone, or soft tissue bulk disease and resection of residual lesions. Patients are followed weekly for 1 month, biweekly for 2 months, monthly for 5 months, and then bimonthly for 1 year.

PROJECTED ACCRUAL: A minimum of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage IV breast carcinoma that is considered incurable by standard treatment Ongoing objective response to prior induction chemotherapy required No brain metastasis Hormone receptor status: Estrogen and progesterone receptor status known

PATIENT CHARACTERISTICS: Age: Over 18 Sex: Not specified Menopausal status: Not specified Performance status: Karnofsky 90-100% Life expectancy: More than 3 months Hematopoietic: Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hemoglobin greater than 9 g/dL Hepatic: Bilirubin less than 1.5 times upper limit of normal (unless due to benign congenital hyperbilirubinemia) PT and aPTT normal Liver biopsy normal if serologic evidence of active hepatitis B or C Renal: Creatinine no greater than 1.2 mg/dL Cardiovascular: No active heart disease LVEF at least 50% and no abnormal wall motion by MUGA scan Pulmonary: DLCO normal Other: Nutritional status adequate (more than 1,000 calories/day orally) HIV negative No other active serious medical or psychiatric disease No other prior malignancy except basal cell skin cancer or carcinoma in situ of the cervix uteri Not pregnant Negative pregnancy test Fertile patients must use effective barrier contraception during and for up to 2 years after study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior mitomycin or nitrosourea No prior anthracycline greater than 500/m2 unless previously received dexrazoxane At least 4 weeks since other prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to pelvis or brain Surgery: At least 2 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1994-02; Primary Completion 2000-12 (Actual); Study Completion 2000-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael DiGiovanna, MD, Study Chair — Yale University
Locations (1):
- Yale Comprehensive Cancer Center, New Haven, Connecticut, United States